CLINICAL TRIAL: NCT05442255
Title: Toxicological Analysis in Chemical Submission
Acronym: TANCS
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP200054; 2019-A03134-53 (Other: ANSM)
Record Dates: First submitted 2022-06-28; First posted 2022-07-01 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Chemical Submission
Keywords: Toxicological analysis; chemical submission; psychoactive substances; date rape drug

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Chemical Submission: Patients with a suspected chemical submission
  Interventions: Other: Toxicological analysis

INTERVENTIONS:
Other: Toxicological analysis — Automated enzymatic assays Automated Immunoassay Urine Screening High Resolution Toxicological Screening

SUMMARY:
The purpose of this study is to carry out a systematic toxicological analysis of all the patients, examined at the UMJ of the Hôtel-Dieu following a complaint for suspected chemical submission. By comparing the toxicological data with the clinical examination data (e.g. treatment intake), the investigators could determine the number of confirmed chemical submissions and the substances involved.

DETAILED DESCRIPTION:
The number of chemical submissions has been constantly increasing in France for several years. The Parisian Center of Evaluation and Information on Pharmacodependence and Addictovigilance collects notifications of chemical submissions demonstrated by toxicological analyses. For the year 2017, 544 notifications were received by this structure. For cases of probable chemical submission, drugs were involved in more than 75% of cases, mostly benzodiazepines. In Europe, there are few cohort studies on the toxicological analysis of suspected chemical submissions. A systematic review of the literature carried out in 2017 by Anderson et al. reports that most studies deal with isolated cases of chemical submission involving a specific and unusual psychoactive substance or are in fact toxicological studies aiming to develop a new analytical technique concerning a substance. Few relevant European cohort studies on this subject have been carried out and most of them are more than ten years old. The Medico-Judicial Unit of the Hôtel-Dieu (UMJ) receives victims of chemical subjection following the filing of a complaint, upon judicial requisition. Complaints can concern a suspicion of chemical submission alone, or a suspicion of chemical submission associated with a suspicion of sexual assault or a robbery. In these cases, the judicial requisition systematically includes a request for toxicological samples (blood and urine). Depending on the data of the investigation, the judicial authority will decide to have the toxicological analyses of these samples performed. In 2018, at the UMJ of Hôtel-Dieu, 231 conservative samples were taken in cases of suspected chemical submissions. As of the writing of this work (November 2019), only 72 samples have been sealed by the judicial authority, i.e. 31.2% of the cases. Moreover, the results of these analyses are not systematically communicated to the UMJ of the Hôtel-Dieu de Paris nor to the patients. Each year, the Medico-Judicial Unit (UMJ) of the Hôtel-Dieu Hospital in Paris receives between 12,000 and 15,000 alleged victims of criminal offences following their filing of a complaint for medical examination on judicial requisition. Among this population, our study will specifically focus on adults who have filed a complaint for suspected chemical submission. The investigators would like to carry out a systematic toxicological analysis of all the patients who have been examined at the UMJ of the Hôtel-Dieu following a complaint for suspected chemical submission. By comparing the toxicological data with the clinical examination data (e.g. treatment intake), the investigators could determine the number of confirmed chemical submissions and the substances involved. This work has several interests. It would allow us to refine our knowledge of the substances used in chemical submissions, and to determine a possible specificity of the substances used in Paris by comparing our data with those existing in the medical literature, at the European and global levels. The data concerning the proven chemical submissions would be transmitted to the CEIP-A, thus allowing an active participation in the toxicovigilance network. A high number of proven chemical submissions would also alert the judicial authorities to the need to carry out toxicological analyses in a more systematic way. Finally, the investigators will systematically propose to the patients included in the study that they receive their results during the follow-up consultation, which is usually carried out within 3 months of the initial consultation. This last point will allow us to improve the management of these patients, by providing them with the answers necessary for the psychological reconstruction process.

ELIGIBILITY:
Inclusion Criteria:

* Be of legal age (≥ 18) on the day of the exam,
* Have filed a complaint for a suspected chemical chemical,
* Be in possession of a judicial requisition requesting the to take biological samples (blood and urine)
* Claim to be the victim of a suspected chemical chemical submission that took place less than 5 days before the consultation,
* Be affiliated or entitled to a social security system,
* Having been informed of the research and not having opposed to his participation.

Exclusion Criteria:

* Patient under court protection
* Minor patient (< 18 ans),
* Patient under guardianship,
* Patient who does not speak French,
* Patient with psychotic / cognitive symptoms that may impair their judgment,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Alleged victims of criminal offences following their filing of a complaint for medical examination on judicial requisition, seen in the Medico-Judicial Unit (UMJ) of the Hôtel-Dieu Hospital in Paris, France.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-07-27 (Actual)

PRIMARY OUTCOMES:
Presence of one or more psychoactive substances | Day of inclusion
  Identify the presence of one or more psychoactive substances in the tests performed (blood).
Presence of one or more psychoactive substances | Day of inclusion
  Identify the presence of one or more psychoactive substances in the tests performed (urines).

SECONDARY OUTCOMES:
Questionnaire | Day of inclusion
  Questionnaire to identify if voluntary intake of one or more psychoactive substance(s) within 24 hours leading to the suspicion of chemical submission.
Quantification of ethanol | Day of inclusion
  Quantification of ethanol and/or ethylglucuronide (its metabolite) in samples
Quantification of ethylglucuronide | Day of inclusion
  Quantification of ethanol and/or ethylglucuronide (its metabolite) in samples

CONTACTS AND LOCATIONS:
Overall Officials: DUFAYET Laurène, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôtel-Dieu Hospital, Paris, IDF, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liautard M, Magny R, Houze P, Deguette C, Alcaraz E, Douaouria S, Gorgiard C, Labat L, Dufayet L. Pro-active drug-facilitated crimes (DFC): a study in the Department of Forensic Medicine of Paris, France. Int J Legal Med. 2024 Mar;138(2):415-430. doi: 10.1007/s00414-023-03090-2. Epub 2023 Sep 28. PMID 37768350